CLINICAL TRIAL: NCT02221219
Title: Indomethacin and Delayed Umbilical Cord Clamp for Preterm Infant IVH
Brief Title: Effects of Delayed Cord Clamp and/or Indomethacin on Preterm Infant Brain Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hong Huang (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Hong Huang, Research Protocol Manager/Clinical/UKHC, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD070792; R01HD070792 (NIH)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Intraventricular Hemorrhage; Periventricular Leukomalacia; Brain Injury; Renal Injury
Keywords: infant; brain injury; renal; indomethacin
MeSH Terms: conditions — Leukomalacia, Periventricular; Brain Injuries | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- immediate cord clamp & placebo IV solution (Placebo Comparator): This Arm will receive immediate clamp of umbilical cord at birth, and an intravenous delivery of placebo drug solution (diluent for active drug, indomethacin) within the first 12hrs of life.
  Interventions: Drug: placebo infusion; Procedure: immediate cord clamp at birth
- delay cord clamp & placebo IV solution (Experimental): A delay in cord clamp for 45 seconds will be instituted in the delivery room. Placebo drug solution will be administered within 12hrs post-birth.
  Interventions: Procedure: delay in umbilical cord clamp at birth; Drug: placebo infusion
- immediate cord clamp & indomethacin IV (Active Comparator): Umbilical cord will be clamped immediately at birth. Indomethacin will be administered IV, starting within 12hrs of life (0.1mg/kg every 24 hrs for three total doses.This intervention is considered 'standard care' at many Neonatology medical facilities. The dose of indomethacin has been shown to be effective in reducing brain bleeds in preterm infants (although there are also data showing safety concerns).
  Interventions: Drug: Indomethacin; Procedure: immediate cord clamp at birth
- indomethacin iv & delayed cord clamp (Experimental): A delay in cord clamp of 45 seconds will be instituted in the delivery room. In addition, indomethacin will be administered iv (initiated within 12hrs of life), 0.1mg/kg every 24 hrs for three total doses.
  Interventions: Drug: Indomethacin; Procedure: delay in umbilical cord clamp at birth

INTERVENTIONS:
Drug: Indomethacin — indomethacin at standard dose for prevention of intraventricular hemorrhage in preterm infants
  Other Names: indocin
  Arms: immediate cord clamp & indomethacin IV; indomethacin iv & delayed cord clamp
Procedure: delay in umbilical cord clamp at birth — provision of a ~45 second delay of umbilical cord clamping at birth in preterm infants (recorded in delivery note)
  Arms: delay cord clamp & placebo IV solution; indomethacin iv & delayed cord clamp
Drug: placebo infusion — saline infusion to match input of indomethacin treatment group (and serve as drug-dosing 'blinding' for bedside staff)
  Arms: delay cord clamp & placebo IV solution; immediate cord clamp & placebo IV solution
Procedure: immediate cord clamp at birth — no delay in umbilical cord clamp; <10sec (recorded in delivery note)
  Arms: immediate cord clamp & indomethacin IV; immediate cord clamp & placebo IV solution

SUMMARY:
Intraventricular hemorrhage (IVH) and periventricular leukomalacia (PVL) are brain lesions that commonly occur in preterm infants and are well-recognized major contributors to long-term brain injury and related disabilities later in life. Despite its prevalence, long term consequences, and enormous medical and social costs, mechanisms of IVH and optimal strategies to prevent or treat its occurrence are poorly defined, especially for extremely premature infants. Only one medical therapy, prophylactic indomethacin during the first 3 days of life, has been shown to prevent or decrease the severity of IVH in preterm infants, but its use is limited by toxic side effects and debatable effects on long-term outcomes. Several small studies and case reports suggest that delayed umbilical cord-clamping (DCC) may also decrease the incidence of IVH in premature infants, but thus far these trials have indomethacin treatment mixed within their cord clamping protocols. The investigators are conducting a randomized, blinded investigation of 4 treatment groups: 1) Control (no intervention); 2) DCC alone; 3) Prophylactic indomethacin alone; 4) Combination of DCC/indomethacin, with respect to survival, IVH or PVL incidence and severity, neurodevelopmental outcomes, and relevant mechanistic effects. With the steady rise in extreme prematurity births and clear links of IVH to long-term disabilities there is a need to improve care for these patients. This multi- disciplinary project addresses an important medical problem for an understudied patient population, where the current practice has clear limitations.

DETAILED DESCRIPTION:
The investigators will compare efficacy and safety of prophylactic indomethacin, DCC, and their combination, in affecting the incidence and severity of IVH/PVL in infants <30wks gestational age (primary outcome measure of 'fraction of survivors with no severe IVH or PVL' among the 4 groups), and longer term neurocognitive function. Other secondary endpoints and investigations include mechanistic effects of prophylactic indomethacin, DCC, and their combination (blood volume/circulatory status, inflammatory stress, progenitor cells) as well as defining relationships between clinical outcomes and mechanistic measurements among treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women admitted >24weeks and <30weeks gestational age,
* in-hospital birth (allowing for cord clamp randomization)

Exclusion Criteria:

* preterm infant <24weeks or >30weeks at birth
* maternal risks identified by obstetrician
* fetal risks identified by obstetrician
* any congenital abnormality of newborn infant
* placental abruption/placental previa
* delivery less than 2hrs from consenting to study participation

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-10-27 (Actual); Study Completion 2021-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Whitehead, RN, Study Director — UK Section of Neonatology; John Bauer, PhD, Principal Investigator — UK Department of Pediatrics; Hong Huang, MD-PhD, Study Director — University of Kentucky Section of Neonatology
Locations (1):
- Kentucky Childrens Hospital Neonatal Intensive Care Unit, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Cord Clamp & Placebo IV Solution | Delay Cord Clamp & Placebo IV Solution | Immediate Cord Clamp & Indomethacin IV | Indomethacin iv & Delayed Cord Clamp
Started | 36 | 87 | 41 | 92
Completed | 36 | 87 | 41 | 92
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Cord Clamp & Placebo IV Solution | Delay Cord Clamp & Placebo IV Solution | Immediate Cord Clamp & Indomethacin IV | Indomethacin iv & Delayed Cord Clamp | Total
Number analyzed (Participants) | 36 | 87 | 41 | 92 | 256
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 26.2 (1.8) | 26.6 (2.0) | 26.6 (1.8) | 26.4 (1.8) | 26.5 (1.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 19 | 47 | 19 | 47 | 132
  Female | 17 | 39 | 21 | 45 | 122
  Unknown | 0 | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 2 | 7
  Not Hispanic or Latino | 32 | 84 | 39 | 90 | 245
  Unknown or Not Reported | 2 | 1 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 10 | 3 | 12 | 31
  White | 27 | 74 | 36 | 76 | 213
  More than one race | 1 | 2 | 1 | 3 | 7
  Unknown or Not Reported | 2 | 1 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 36 | 87 | 41 | 92 | 256
Birth Weight [Mean (Standard Deviation); unit: grams] | 797.2 (267.4) | 935.1 (295.0) | 902.4 (369.8) | 916.8 (254.8) | 903.9 (291.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Survivors With no Severe IVH (Grades 3 or 4) or PVL
Description: determined by head ultrasound in Neonatal Intensive Care Unit (NICU) and single head MRI at 38weeks corrected gestational age
Time Frame: within first 60 days of life
Measure: Number; unit: percent of participants
Arm/Group | Immediate Cord Clamp & Placebo IV Solution | Delay Cord Clamp & Placebo IV Solution | Immediate Cord Clamp & Indomethacin IV | Indomethacin iv & Delayed Cord Clamp
Number analyzed (Participants) | 36 | 87 | 41 | 92
percent of participants | 22.2 | 14.9 | 17.1 | 10.9

2. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: measures of serum creatinine and urine output during Neonatal Intensive Care Unit (NICU) stay. General measures of renal injury (which is a common risk of indomethacin treatment in this patient population).
Time Frame: first 60 days of life
Measure: Number; unit: participants
Arm/Group | Immediate Cord Clamp & Placebo IV Solution | Delay Cord Clamp & Placebo IV Solution | Immediate Cord Clamp & Indomethacin IV | Indomethacin iv & Delayed Cord Clamp
Number analyzed (Participants) | 36 | 87 | 41 | 92
participants
  No acute kidney injury | 20 | 48 | 23 | 48
  Grade 1 Acute Kidney Injury | 8 | 27 | 15 | 29
  Grade 2 Acute Kidney Injury | 6 | 8 | 3 | 14
  Grade 3 Acute Kidney Injury | 2 | 4 | 0 | 1
  Grade 4 Acute Kidney Injury | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Hematological Status
Description: hematocrit, ferritin, hemoglobin at various times during NICU stay
Time Frame: first 60 days of life
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Inflammatory Stress
Description: measurement of inflammatory biomarkers (CRP, Interleukin-6, soluble ICAM) at various times during NICU stay
Time Frame: first 60 days of life
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Circulating Progenitor Cell Subpopulations
Description: measures of several progenitor cell subtypes in blood during the NICU stay
Time Frame: first 60 days of life
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Neurocognitive Assessments at Post-NICU Followup
Description: standardized neurocognitive assessments done at NICU graduate clinic.
Time Frame: up to 24 months of corrected gestational age
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: First 60 days of life.
Arm/Group | Immediate Cord Clamp & Placebo IV Solution | Delay Cord Clamp & Placebo IV Solution | Immediate Cord Clamp & Indomethacin IV | Indomethacin iv & Delayed Cord Clamp
All-Cause Mortality (participants affected / at risk) | 6/36 | 10/87 | 2/41 | 6/92
Serious Adverse Events (participants affected / at risk) | 5/36 | 7/87 | 3/41 | 10/92
Other Adverse Events (participants affected / at risk) | 0/36 | 0/87 | 0/41 | 0/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Cord Clamp & Placebo IV Solution (N=36) | Delay Cord Clamp & Placebo IV Solution (N=87) | Immediate Cord Clamp & Indomethacin IV (N=41) | Indomethacin iv & Delayed Cord Clamp (N=92)
Necrotizing Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extreme Prematurity (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 5 (5) | 1 (1) | 5 (5)
Free Air in Abdomen (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Septic Shock (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bowel Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
CMV (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiorgan Failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT02221219/Prot_SAP_ICF_000.pdf